CLINICAL TRIAL: NCT03999801
Title: A Long-term Follow-Up Study to Evaluate the Safety and Efficacy of RGX-314 Following Subretinal Administration in Participants With Neovascular Age-related Macular Degeneration and Fellow Eye Treatment Substudy
Brief Title: Long-term Follow-Up Study of RGX-314 and Fellow Eye Substudy
Acronym: RGX-314 SRLTFU
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGX-314-5101
Record Dates: First submitted 2019-06-18; First posted 2019-06-27 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Neovascular Age-related Macular Degeneration; Wet Macular Degeneration
Keywords: gene therapy; wet AMD; nAMD
MeSH Terms: conditions — Wet Macular Degeneration

STUDY DESIGN:
Intervention Model Description: 1 main Observational study arm, 1 RGX-314 Fellow Eye Treatment substudy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Main Observational Study (No Intervention): All subjects that previously received RGX-314 in a subretinal administration parent study are enrolled into this arm.
- RGX-314 Fellow Eye Treatment Substudy (Experimental): RGX-314 Fellow Eye Treatment
  Interventions: Genetic: RGX-314

INTERVENTIONS:
Genetic: RGX-314 — AAV8 vector containing a transgene for anti-VEGF Fab
  Arms: RGX-314 Fellow Eye Treatment Substudy

SUMMARY:
This is a prospective, observational study designed to evaluate the long-term safety and efficacy of RGX-314. Eligible participants are those who were previously enrolled in a clinical study in which they received a single subretinal administration of RGX-314 in their study eye. Enrollment of each participant in the current study should occur after the participant has completed either the end of study or early termination visit in the previous (parent) clinical study. Participants will be followed for up to 5 years post-RGX-314 administration (inclusive of the parent study). After enrollment and a 6-month follow-up visit, participants will attend at least annual study visits through the end of the 5-year post-RGX-314 administration follow-up period.

Additionally, an interventional fellow eye treatment substudy will evaluate the safety, efficacy, and immunogenicity of subretinal RGX-314 administration in the fellow eye of participants having bilateral disease who previously received a subretinal injection of RGX-314 in their study eye. Participants who qualify for the substudy will receive subretinal administration of RGX-314 in their fellow eye and complete 13 study visits in a 54-week period. Following completion of the substudy participants will continue in the observational portion of the study for up to 5 years post RGX-314 administration in their fellow eye.

ELIGIBILITY:
Main Observational Study:

Inclusion Criteria:

1. Able and willing to provide written consent
2. Previously enrolled in a clinical study of RGX-314 and received a single subretinal administration of RGX-314

Exclusions Criteria:

1. None

Fellow Eye Substudy:

Inclusion Criteria

1. Age ≤ 93 years
2. Currently or previously enrolled in the main observational study
3. Diagnosis of bilateral choroidal neovascularization secondary to age-related macular degeneration
4. Active nAMD in the fellow eye
5. BCVA between ≤ 80 and ≥ 20 letters in the fellow eye

Exclusion Criteria:

1. CNV or macular edema in the fellow eye secondary to causes other than nAMD
2. Subfoveal fibrosis or atrophy in the fellow eye
3. Advanced glaucoma or history of secondary glaucoma in the fellow eye or any invasive procedure to treat glaucoma
4. Myocardial infarction, cerebrovascular accident, or transient ischemic attack within the past 6 months
5. History of intraocular surgery in the fellow eye within 12 weeks of screening
6. History of intravitreal therapy, such as intravitreal steroid injection or investigational product, other than an intravitreal therapy for nAMD, in the fellow eye within 6 months of screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 865 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular adverse events and any serious adverse events in the study eye | 5 years inclusive of parent study
Fellow eye substudy: Incidence of ocular adverse events and any serious adverse events in the fellow eye | 54 weeks

SECONDARY OUTCOMES:
Change from baseline in best corrected visual acuity (BCVA) in the study eye | 5 years inclusive of parent study
  Mean change and proportion of participants losing greater than or equal to 5, 10, and 15 letters
Change from baseline in Central Retinal Thickness (CRT) in the study eye | 5 years inclusive of parent study
  Mean change from baseline in CRT as measured by spectral domain optical coherence tomography (SD-OCT)
Number of supplemental anti-VEGF injections in the study eye | 5 years inclusive of parent study
  Mean number of supplemental anti-VEGF injections based on chart review
Number of retinal specialist visits for the study eye | 5 years inclusive of parent study
  Mean number of retinal specialist visits attended for nAMD based on chart review
Fellow eye substudy: Change from baseline in best corrected visual acuity | 54 weeks
  Mean change from baseline in BCVA in the fellow eye
Fellow eye substudy: Change from baseline in Central Retinal Thickness in the fellow eye | 54 weeks
  Mean change from baseline in CRT in the fellow eye as measured by SD-OCT
Fellow eye substudy: Number of supplemental anti-VEGF injections in the fellow eye | 54 weeks
  Mean number of supplemental anti-VEGF injections in the fellow eye
Fellow eye substudy: Aqueous and Serum RGX-314 transgene product (TP) concentrations in the fellow eye | 54 weeks
  Fellow eye aqueous and serum RGX-314 TP concentrations at assessed time points
Fellow eye substudy: Immunogenicity measurements in the fellow eye | 54 weeks
  Fellow eye immunogenicity measurements at assessed timepoints

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Retinal Research Institute, LCC, Phoenix, Arizona
  - California Retina Consultants CRC, Santa Barbara, California
  - Johns Hopkins University, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Sierra Eye Associates, Reno, Nevada
  - University of Pennsylvania Department of Ophthalmology, Philadelphia, Pennsylvania
  - MidAtlantic Retina, Philadelphia, Pennsylvania
  - Charles Retina Institute, Germantown, Tennessee
  - Retina Consultants of Texas Research Center, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No